CLINICAL TRIAL: NCT02069405
Title: Relaxation Music to Lower Heart Rate Prior to Cardiac CT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 13-6798-AE
Record Dates: First submitted 2013-12-11; First posted 2014-02-24 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2013-12

CONDITIONS: Coronary Artery Disease and Cardiac Anatomy; Patients Undergoing Coronary CT Angiogram; Patients Undergoing CT Pulmonary Vein Angiogram; Patients Undergoing CT Calcium Score
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music Group plus normal standard of care (Experimental): Patients will listen to music prior and during the scan
  Interventions: Other: Relaxation Music
- Control Group - Normal standard of care (No Intervention)

INTERVENTIONS:
Other: Relaxation Music
  Arms: Music Group plus normal standard of care

SUMMARY:
To acquire low radiation dose and good quality cardiac CT images requires scanning at low heart rates which is usually done with beta-blockers. However, in some patients beta-blockers have little effect. This is thought to be due to a different mechanism of action which continues to maintain the heart rate despite administration of beta-blockers. This study aims to look at the effect of music or relaxation tracks to reduce patient heart rate as anxiety is thought to play a role in maintaining high heart rates. This study will randomise patients into a normal standard of care group compared to a normal standard of care group with music/ relaxation track and compare heart rate, radiation dose, image quality, amount of beta-blocker used and patient experience via a State-Trait Anxiety Inventory (STAI) questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 years and above
* All patients coming in for non-contrast enhanced calcium score CT, pulmonary vein angiogram, or coronary CT Angiogram

Exclusion Criteria:

* Deaf
* CT for Transcatheter aortic valve implantation (TAVI) or congenital heart disease patients
* Poor english literacy
* Pacemaker
* Post CABG
* Post heart transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate | Same day as CT scan
  Unit of measure - beats per minute

SECONDARY OUTCOMES:
Radiation Dose | Same day as CT scan
  Unit of measure - millisieverts
Image Quality | Same day as CT scan
  Measurement tool - Likert Scale. Review of images by two highly experienced cardiac radiologists
IV metoprolol dose | Same day as CT scan
  Unit of measurement - milligrams
Patient Satisfaction | Same day as CT scan
  Measurement tool - Modified state-trait anxiety inventory (STAI) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Elsie Nguyen, MD, Principal Investigator — University Health Network, Joint Department of Medical Imaging; Ming-Yen Ng, BMBS, Study Chair — University Health Network, Joint Department of Medical Imaging
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada